CLINICAL TRIAL: NCT03756467
Title: Girl Empower: Studying the Impact of Mentorship, Asset Building, Caregiver Discussion Groups, and Cash Transfers on Reducing Girl's Vulnerability to Sexual Exploitation and Abuse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Population Council (Other)
Collaborators: World Bank (Other); International Rescue Committee (Other); City University of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 645
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Adolescent Behavior; Sexual Violence
Keywords: Adolescent Behavior; Sexual Violence
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: The impact evaluation study is a cluster-randomized controlled trial among 100 communities with three study arms: control (no intervention), GE, and GE+.
Who Masked: Participant
Masking Description: The impact evaluation is a cluster-randomized controlled trial with three study arms: control (no program), GE, and GE+. GE refers to the Girl Empower program alone, while GE+ adds small cash transfers to the families of eligible girls as an incentive to increase take-up of GE attendance in weekly sessions. The study team will conduct a baseline survey of all girls age 13-14 and their caregiver in 100 communities in Nimba County, Liberia. Communities will then be randomized, blocking on number of girl in the community and % of girls enrolled in school, to one of the 3 study arms. Two years following the baseline survey (1 year following program completion), the study team will conduct an endline survey in all 100 communities with the same girls and caregivers and compare outcomes in the three study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (No Intervention): 1) the Girl Empower life skills curriculum, facilitated by local mentors; 2) caregiver discussion group, facilitated by IRC staff
- Arm 2 (Experimental): 1) the Girl Empower life skills curriculum, facilitated by local mentors; 2) caregiver discussion group, facilitated by IRC staff; and 3) savings account start-up
  Interventions: Behavioral: Girl Empower Program
- Arm 3 (Active Comparator): 1) the Girl Empower life skills curriculum, facilitated by local mentors; 2) caregiver discussion group, facilitated by IRC staff; and 3) savings account start-up.
  Interventions: Behavioral: Girl Empower Program

INTERVENTIONS:
Behavioral: Girl Empower Program — Girl Empower (GE) encourages adolescent girls living in rural areas of Nimba County, Liberia to partake in weekly mentored community-based workshops on life skills, selfcare, and financial literacy.
  Arms: Arm 2; Arm 3

SUMMARY:
Girl Empower (GE) is a program designed to equip girls with the skills and experiences necessary to make healthy, strategic life choices and to stay safe from sexual exploitation and abuse.

DETAILED DESCRIPTION:
The GE program is unique in its approach because it addresses girls' needs holistically. The girls' activities will take place in girl-only safe spaces located in their communities and contains the following components: Mentorship: girls have access to older female mentors. Mentors both provide weekly group-based and one-to-one interaction with girls as well as teach them critical skills; Asset building: Girls will have access to life skills and financial literacy training. This includes setting up savings accounts so girls practice their financial literacy skills, Monthly caregiver discussion groups among guardians of program girls, Capacity building and training of local health and psychosocial service providers to provide quality services to survivors of gender-based violence Intervention communities will either receive the GE program alone or the GE program with the plus small cash transfers to the girls' families as an incentive to attendance in weekly sessions (GE+).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, eligible girls aged 13 to 14 years of age.

Exclusion Criteria:

-

Ages: 13 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2200 (Estimated)
Dates: Start 2017-07-12 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Sexual Violence Index | 40 weeks
  The primary outcome of interest is an index of sexual violence at the individual level.
  The index is composed of four questions in the endline survey instrument. The construction of the index, and a detailed description of its components is described in the pre-analysis plan (PAP) document uploaded under the "Analysis Plan" in this registration.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Hallman, Ph.D., Principal Investigator — Population Council
Locations (1):
- University of Liberia, Monrovia, Liberia

IPD SHARING:
Plan to Share IPD: No